CLINICAL TRIAL: NCT01081405
Title: Allogeneic Hematopoietic Cell Transplantation Using a Non-myeloablative Preparative Regimen of Total Lymphoid Irradiation and Anti-Thymocyte Globulin for Patients With Hematologic Malignancies
Brief Title: Total Lymphoid Irradiation and Anti-Thymocyte Globulin in the Allogeneic Hematopoietic Cell Transplantation
Acronym: TLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLI-001-2007; 2007-005563-10 (EudraCT Number)
Record Dates: First submitted 2010-03-02; First posted 2010-03-05 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: HEMATOLOGIC MALIGNANCIES
Keywords: ALLOGENEIC HEMATOPOIETIC CELL TRANSPLANTATION; TOTAL LYMPHOID IRRADIATION; ANTI-THYMOCYTE GLOBULIN
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TOTAL LYMPHOID IRRADIATION (Experimental): Allogeneic Hematopoietic Cell Transplantation Using a Non-myeloablative Preparative Regimen of Total Lymphoid Irradiation and Anti-Thymocyte Globulin for Patients with Hematologic Malignancies
  Interventions: Other: TOTAL LYMPHOID IRRADIATION

INTERVENTIONS:
Other: TOTAL LYMPHOID IRRADIATION — Allogeneic Hematopoietic Cell Transplantation Using a Non-myeloablative Preparative Regimen of Total Lymphoid Irradiation and Anti-Thymocyte Globulin for Patients with Hematologic Malignancies

SUMMARY:
To exploit the curative potential of allografting, the ultimate clinical goal is to separate GVL from GVHD. In murine preclinical models, recipients of allogeneic hematopoietic cell transplants after a preparative regimen of total lymphoid irradiation (TLI) and antithymocyte globulin (ATG) did not develop GVHD. The murine TLI/ATG study was turned into a clinical phase I protocol for patients with hematological malignancies, and a reduction of acute GVHD to < 3% was observed (Lowsky R et al, N Engl J Med). This suggests that specific immune mechanisms control GVHD and preserve GVL. The study will include patients with lympho and myeloproliferative diseases. The conditioning regimen will consist of TLI [ten 80 cGy fractions on day -11 through day -7 and on day -4 through day -1; the radiation field (four fields-two anterior and two posterior) involves all major lymphoid organs including the thymus, spleen and lymph nodes] and ATG (five i.v. doses at 1.5 mg/kg/day from day -11 through day -7). G-CSF mobilised hematopoietic cells, collected on days -1 and 0, from HLA-identical siblings or unrelated donors will be infused on day 0. Post-transplant immunosuppression will consist of oral cyclosporine (at 6.25 mg/kg/d) from day -3 and micophenolate mophetile (at 15 mg/Kg bid) from day +1. The clinical primary objective is to reduce the incidence of GVHD to < 5%, with better survival and quality of life.

DETAILED DESCRIPTION:
PATIENT ENROLMENT.

It is expected that about 15 patients / year will be enrolled in this phase I-II protocol. Patient selection will be based on the following criteria:

Eligibility Criteria:

1. Any patient with one of the following lympho or myeloproliferative malignancies or syndromes in whom allogeneic NST is warranted. Patients with other selected malignancies/disorders may also be considered but must be approved by the transplant team and the Principal Investigator.
2. Patient age > 50 years, or for patients <50 years of age but because of pre-existing medical conditions or prior therapy are considered to be at high risk for regimen-related toxicity associated with conventional myeloablative transplants.
3. an HLA-identical sibling or matched unrelated donor is available. Patients with one antigen mismatched donors can be considered but only after discussion with the transplant team and the Principal Investigator.

STEM CELL TRANSPLANTATION:

(A) TLI Administration: see "brief description" (B) ATG: Thymoglobulin will be administered five times intravenously at 1.5 mg/kg/day from day -11 through day -7 for a total dose of 7.5 mg/kg. Thymoglobulin doses will be based on the adjusted ideal body weight. Premedication for thymoglobulin will include solumedrol 1.0 mg/kg.

Mobilized PBPC: The minimum cell doses (based on recipient body weight) for transplants are > 5x106 CD34+ cells/kg. Cells collected on days -1 and 0 will be pooled and processed for infusion on day 0. Fresh cells (not frozen) are to be infused. For related donor transplants, if the target cell dose is not achieved then a third apheresis procedure may be performed on day+1 and the cells infused on the same day. Collection of cells for unrelated donor transplants will be coordinated through the Italian bone Marrow Transplant Registry and subject to the rules of that Program. If mobilized PBPC is not available through certain collection centers then bone marrow will be used.

(F) Cyclosporine (CSP): CSP is given at 6.25 mg/kg p.o. b.i.d (9 a.m and 9 p.m.) from day -3 until after the day +56 chimerism results are obtained. CSP will be tapered after the day +56 chimerism results are obtained. If the day +56 chimerism results show >40% donor cells in the CD3+ lineage, and the patient is without evidence of GVHD then CSP taper will begin. The CSP will be tapered at 6% every week. Modifications of the taper schedule may be indicated if significant disease progression occurs early post-transplantation or the patient develops GVHD.

(G) Mycophenylate mofetil (MMF): Administration of MMF will begin at 15 mg/kg po on day 0, at 5-10 hours after mobilized PBPC infusion is complete. Thereafter,beginning on day +1 MMF is taken at 15 mg/kg po b.i.d. (30 mg/kg/day) if transplantation was using a matched related donor and 15 mg/kg po t.i.d if from a matched unrelated donor or a one antigen mismatched donor. Doses will be rounded up to the nearest 250 mg (capsules are 250 mg). MMF will be stopped on day +28 for matched related donors and for one antigen mismatched or unrelated donors beginning day +40 MMF will be tapered by 10% weekly till off, typically by day +96.

POST-TRANSPLANT FOLLOW-UP

Clinical: The incidence, severity and extent of acute and chronic GVHD will be monitored and scored according to standard criteria. As well, documented and presumed post-transplant infectious complications, rate of relapse, event-free and overall survival and transplant related mortality will be recorded.

Assessment of Disease Response: Since the diseases treated on this protocol are heterogenous, appropriate disease specific studies will be performed to evaluate response to transplant. Responses will be classified as continued complete remission (CCR), achieved complete remission (CRa), partial response (PR), progressive disease (PD), or no response (NR). Disease response will be according to accepted criteria. All cases of progressive disease should be discussed with the Principal Investigators. If patients show evidence of progressive disease then they may be candidates for donor lymphocyte infusion.

ELIGIBILITY:
Inclusion Criteria:

(A) Any patient with one of the following hematolymphoid malignancies or syndromes in whom allogeneic NST is warranted. Specific disease categories include: indolent advanced stage Non-Hodgkin Lymphomas, Mantle Cell Lymphoma, Chronic Lymphocytic Leukemia, Hodgkin Disease, Acute Leukemias in any complete remission, Aplastic Anemia, Paroxsymal Nocturnal Hemoglobinuria, Myelodysplastic and Chronic Myeloproliferative Syndromes, Multiple Myeloma. Patients with other selected malignancies/disorders may also be considered but must be approved by the transplant team and the Principal Investigator.

(B) Elderly patients age > 50 < 70 years, or for patients <50 years of age but because of pre-existing medical conditions or prior therapy are considered to be at high risk for regimen-related toxicity associated with conventional myeloablative transplants, or because of refusal to undergo conventional myeloablative regimes.

(C) A fully HLA-identical sibling or matched unrelated donor is available. Patients with one antigen mismatched donors can be considered but only after discussion with the transplant team and the Principal Investigator.

(D) Patient must be competent to give consent.

Exclusion Criteria:

(A) Patients with progressive hematolymphoid malignancies despite conventional therapies, or acute leukemias not in complete remission.

(B) Uncontrolled CNS involvement with disease

(C) Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment

(D) Females who are pregnant

(E) Organ dysfunction defined as follows:

* Cardiac function: ejection fraction <30% or uncontrolled cardiac failure
* Pulmonary: DLCO <40% predicted
* Liver function abnormalities: elevation of bilirubin to > 3 mg/dl and/or transaminases >4x the upper limit of normal
* Renal: creatinine clearance <50 cc/min (24 hour urine collection)

(F) Karnofsky performance score < 60%

(G) Patients with poorly controlled hypertension on multiple antihypertensives

(H) Documented fungal disease that is progressive despite treatment

(I) Viral infections: HIV positive patients. Hepatitis B and C positive patients will be evaluated on a case by case basis

(J) Psychiatric disorders or psychosocial problems which in the opinion of the primary physician or Principal Investigator would place the patient at unacceptable risk from this regimen.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure not applicable | Not reached

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U. Città della Salute e della Scienza di Torino, Torino, Italy